CLINICAL TRIAL: NCT00513409
Title: Phase II, Observer-blind Follow-up Study to Assess reacto-and Immunogenicity of GSK Biologicals' Pneumococcal Conjugate Vaccine (GSK1024850A), When Given as Booster in Primed Children or as 2-dose Catch-up in Unprimed Children.
Brief Title: Assess Reacto- and Immunogenicity of Pneumococcal Conjugate Vaccine When Given as Booster or a 2 Dose Catch up Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110031
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-05

CONDITIONS: Infections, Streptococcal
Keywords: Immunogenicity; Pneumococcal disease; Safety; Booster vaccination; Pneumococcal vaccine
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Care Provider, Investigator

ARMS (2):
- Synflorix Booster Group (Experimental): Subjects previously primed with Synflorix™ and receiving in the current study Havrix™ co-administered with Infanrix™ hexa (Dose 1) and Synflorix™ (Dose 2).
  Interventions: Biological: Synflorix; Biological: Infanrix Hexa; Biological: Havrix
- Synflorix Catch-up Group (Experimental): Subjects previously primed with Havrix™ co-administered with Infanrix™ hexa and receiving in the current study Synflorix™ co-administered with Infanrix™ hexa (Dose 1) and Synflorix™ (Dose 2).
  Interventions: Biological: Synflorix; Biological: Infanrix Hexa

INTERVENTIONS:
Biological: Synflorix — Intramuscular injection, 1 or 2 doses
Biological: Infanrix Hexa — 1 Intramuscular injection
  Other Names: DTPa-HBV-IPV/Hib
Biological: Havrix — 1 Intramuscular injection
  Arms: Synflorix Booster Group

SUMMARY:
This is a booster study in 2 groups of healthy children less than 3 years old to measure the reactogenicity, safety and immunogenicity of GSK Biologicals' pneumococcal conjugate vaccine, when given as a booster or as a two-dose catch-up vaccination.

This protocol posting deals with objectives and outcome measures of the booster phase. The objectives and outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00338351).

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 18-21 months of age at the time of vaccination.
* Subjects who previously participated in the primary study and received 3 doses of study or control vaccines during the primary study.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the booster doses of study vaccines, or planned use during the study period (active phase and extended safety follow-up).
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month (30 days) before the booster doses of vaccine(s) and during the active phase of the study (up to the follow-up visit (Visit 3)).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures (subjects who have had a single, uncomplicated febrile convulsion in the past can be included) or progressive neurological disease.
* Acute disease at the time of enrolment.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the booster doses of study vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products within the last 3 months prior to booster or follow-up vaccination or planned administration during the active phase of the study.

Ages: 18 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2007-08-22; Primary Completion 2008-02-20 (Actual); Study Completion 2008-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lagos RE, Munoz AE, Levine MM, Lepetic A, Francois N, Yarzabal JP, Schuerman L. Safety and immunogenicity of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Chilean children. Hum Vaccin. 2011 May;7(5):511-22. doi: 10.4161/hv.7.5.14634. Epub 2011 May 1. PMID 21441782
- [Background] Lagos R et al. 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHiD-CV) given as booster dose or 2-dose catch-up in Chilean children. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110031 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110031 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110031 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110031 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110031 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110031 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Started | 84 | 79
Completed | 82 | 73
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Visit 3 not done | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group | Total
Number analyzed (Participants) | 84 | 79 | 163
Age, Continuous [Mean (Standard Deviation); unit: Months] | 18.3 (0.44) | 18.3 (0.50) | 18.3 (0.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 44 | 83
  Male | 45 | 35 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Grade 3 Symptoms (Solicited and Unsolicited)
Description: Grade 3 symptoms are symptoms which prevent normal, everyday activities (e.g. in a young child such symptom would prevent attendance at school/ kindergarten/ a day-care center and would cause the parents/guardians to seek medical advice).
Time Frame: Within 4 days after the administration of any study vaccine dose
Population: Analysis was performed on all subjects included in the Total Vaccinated Cohort, who returned the symptom sheet.
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 84 | 78
subjects
  Any symptoms | 32 | 36
  General symptoms | 6 | 14
  Local symptoms | 30 | 32

2. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: Within 4 days after the administration of any study vaccine dose
Population: Analysis was performed on all subjects included in the Total Vaccinated Cohort, who returned the symptom sheet.
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 84 | 78
subjects
  Pain | 57 | 63
  Redness | 49 | 52
  Swelling | 44 | 47

3. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever, irritability and loss of appetite.
  Fever was defined as rectal temperature ≥ 38 degrees Celsius.
Time Frame: Within 4 days after the administration of any study vaccine dose
Population: Analysis was performed on all subjects included in the Total Vaccinated Cohort, who returned the symptom sheet.
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 84 | 78
subjects
  Drowsiness | 33 | 36
  Fever | 30 | 40
  Irritability | 56 | 55
  Loss of appetite | 35 | 37

4. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 31 days after the administration of any study vaccine dose
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 84 | 79
subjects | 47 | 47

5. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events During the Active Phase of the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Throughout the active phase of the study ( from the beginning of the booster phase up to 1 month after the second booster dose)
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 84 | 79
subjects | 1 | 0

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events Throughout the Entire Study Period
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Throughout the entire study period (from the beginning of the booster phase up to the end of the 6-month extended safety follow-up)
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 84 | 79
subjects | 1 | 0

7. Secondary Outcome: Number of Subjects With Vaccine Pneumococcal Serotype Antibody Concentrations Above the Cut-off Value
Description: Anti-pneumococcal antibody cut-off value assessed was 0.20 microgram per milliliter (μg/mL).
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F.
Time Frame: Before (pre) and one month after (post) the administration of Dose 2
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 80 | 73
subjects
  Anti-1 Pre (N=79; 72) | 43 | 1
  Anti-1 Post (N=78; 70) | 78 | 70
  Anti-4 Pre (N=75; 73) | 45 | 3
  Anti-4 Post (N=77; 70) | 77 | 70
  Anti-5 Pre (N=76; 70) | 58 | 7
  Anti-5 Post (N=78; 70) | 77 | 70
  Anti-6A Pre (N=76; 72) | 66 | 36
  Anti-6A Post (N=77; 70) | 71 | 64
  Anti-6B Pre (N=76; 73) | 55 | 1
  Anti-6B Post (N=78; 70) | 76 | 59
  Anti-7F Pre (N=70; 68) | 60 | 8
  Anti-7F Post (N=78; 70) | 77 | 70
  Anti-9V Pre (N=78; 72) | 71 | 6
  Anti-9V Post (N=79; 70) | 79 | 69
  Anti-14 Pre (N=76; 71) | 69 | 20
  Anti-14 Post (N=79; 70) | 79 | 70
  Anti-18C Pre (N=77; 73) | 68 | 5
  Anti-18C Post (N=78; 70) | 78 | 70
  Anti-19A Pre (N=78; 73) | 72 | 50
  Anti-19A Post (N=78; 70) | 78 | 70
  Anti-19F Pre (N=80; 72) | 76 | 19
  Anti-19F Post (N=78; 70) | 78 | 70
  Anti-23F Pre (N=76; 71) | 59 | 3
  Anti-23F Post (N=78; 70) | 78 | 66

8. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes Above the Cut-off Value
Description: Cut-off value for opsonophagocytic activity against pneumococcal antibody assessed was ≥ 8
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F.
Time Frame: Before (pre) and one month after (post) the administration of Dose 2
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity,on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 29 | 28
subjects
  Opsono-1 Pre (N=28; 25) | 12 | 1
  Opsono-1 Post (N=25; 25) | 25 | 13
  Opsono-4 Pre (N=17; 19) | 7 | 1
  Opsono-4 Post (N=24; 18) | 24 | 18
  Opsono-5 Pre (N=19; 23) | 13 | 1
  Opsono-5 Post (N=20; 25) | 20 | 21
  Opsono-6A Pre (N=20; 25) | 12 | 2
  Opsono-6A Post (N=19; 19) | 14 | 12
  Opsono-6B Pre (N=22; 25) | 12 | 3
  Opsono-6B Post (N=24; 27) | 22 | 13
  Opsono-7F Pre (N=17; 12) | 16 | 4
  Opsono-7F Post (N=25; 26) | 25 | 26
  Opsono-9V Pre (N=20; 17) | 20 | 11
  Opsono-9V Post (N=23; 23) | 23 | 22
  Opsono-14 Pre (N=16; 11) | 14 | 5
  Opsono-14 Post (N=21; 25) | 21 | 25
  Opsono-18C Pre (N=29; 28) | 12 | 3
  Opsono-18C Post (N=26; 27) | 25 | 27
  Opsono-19A Pre (N=18; 18) | 0 | 0
  Opsono-19A Post (N=23; 19) | 14 | 5
  Opsono-19F Pre (N=22; 23) | 17 | 2
  Opsono-19F Post (N=20; 21) | 20 | 20
  Opsono-23F Pre (N=21; 16) | 18 | 8
  Opsono-23F Post (N=25; 25) | 25 | 25

9. Secondary Outcome: Number of Subjects With Anti-protein D Antibody Concentrations Above the Cut-off Value
Description: Anti-protein D antibody cut-off value assessed was ≥ 100 Enzyme-Linked Immuno Sorbent Assay (ELISA) unit per milliliter (EL.U/mL).
Time Frame: Before (pre) and one month after (post) the administration of Dose 2
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity,on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 77 | 70
subjects
  Pre (N= 73; 69) | 72 | 44
  Post (N= 77; 70) | 77 | 70

10. Secondary Outcome: Anti-hepatitis A Virus Antibodies Concentration
Description: Concentration of anti-hepatitis A antibodies given as geometric mean concentration (GMC) in milli-international units per milliliter (mIU/mL).
Time Frame: Before (pre) and one month after (post) the administration of Dose 2
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity,on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 19 | 21
mIU/mL
  Pre (N=18; 21) | 30.3 [16.3 to 56.3] | 539.9 [231.0 to 1261.9]
  Post (N=19; 19) | 495.5 [228.0 to 1076.7] | 478.5 [199.4 to 1148.2]

11. Secondary Outcome: Number of Subjects With Anti-hepatitis A Antibody Concentrations Above the Cut-off Value
Description: Anti-hepatitis A antibodies cut-off value assessed was ≥ 15 mIU/mL.
Time Frame: Before (pre) and one month after (post) the administration of Dose 2
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Number analyzed (Participants) | 19 | 21
subjects
  Pre (N=18; 21) | 12 | 21
  Post (N=19; 19) | 18 | 19

ADVERSE EVENTS:
Arm/Group | Synflorix Booster Group | Synflorix Catch-up Group
Serious Adverse Events (participants affected / at risk) | 1/84 | 0/79
Other Adverse Events (participants affected / at risk) | 78/84 | 75/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Booster Group (N=84) | Synflorix Catch-up Group (N=79)
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Booster Group (N=84) | Synflorix Catch-up Group (N=79)
Bronchitis (Infections and infestations) | 15 | 16
Nasopharyngitis (Infections and infestations) | 6 | 14
Diarrhoea (Gastrointestinal disorders) | 6 | 8
Injection site induration (General disorders) | 7 | 7
Rhinitis (Infections and infestations) | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 2
Pain (General disorders) | 57 | 63
Redness (General disorders) | 49 | 52
Swelling (General disorders) | 44 | 47
Drowsiness (General disorders) | 33 | 36
Fever (Rectally) (General disorders) | 30 | 40
Irritability (General disorders) | 56 | 55
Loss of appetite (General disorders) | 35 | 37
Pharyngitis (Infections and infestations) | 6 | 8
Pyrexia (General disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.